CLINICAL TRIAL: NCT06427993
Title: Urine Exfoliated Cell DNA Methylation Detection for Urothelial Carcinomas Diagnosis in Patients With Hematuria--A Prospective, Single-center, Cohort Study
Brief Title: Urine DNA Methylation Detection for Hematuria Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CH_Hematuria_Metest
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Hematuria; Urothelial Carcinoma; Bladder Cancer; Ureter Cancer; Renal Pelvis Cancer
Keywords: Hematuria; Urothelial Carcinoma; Urine DNA Methylation
MeSH Terms: conditions — Hematuria; Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine sediment DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Hematuria, a common symptom of urinary system diseases, can result from various causes including infection, stones, trauma, and tumors. Urothelial carcinoma (UC), the most common malignancy of the urinary system, often presents with hematuria. Current diagnostic methods like urine cytology and cystoscopy have limitations in sensitivity and specificity, and cystoscopy is invasive. DNA methylation biomarkers offer potential for non-invasive UC detection, improving diagnostic accuracy in hematuria patients.

Objective: This study aims to evaluate the diagnostic performance of DNA methylation biomarkers in detecting UC in patients with hematuria.

Methods: This prospective pilot study will involve collecting preoperative urine samples from hematuria patients for DNA methylation testing using MSRE-qPCR. Sample size calculation was based on an assumed 25% prevalence of UC in hematuria patients, resulting in a total of 71 participants after accounting for a 20% dropout rate. Sensitivity, specificity, and diagnostic performance will be assessed using ROC curves.

Conclusion: This study seeks to validate the effectiveness of urine DNA methylation testing for UC detection in hematuria patients, providing a basis for its clinical application and informing the design of larger future studies.

DETAILED DESCRIPTION:
1. Background Hematuria is a common symptom of urinary system diseases and can be caused by various factors, including infection, stones, trauma, and tumors. Urothelial carcinoma (UC) is the most common malignant tumor of the urinary system, primarily occurring in the bladder, renal pelvis, and ureter. The early symptoms of UC are often not obvious, with hematuria being the most common symptom. However, current diagnostic methods such as urine cytology and cystoscopy have limitations in sensitivity and specificity for diagnosing UC. Additionally, cystoscopy is invasive and can cause discomfort for patients. DNA methylation biomarkers have shown potential in detecting UC, providing a non-invasive method to improve diagnostic sensitivity and specificity, especially in patients with hematuria.
2. Objective This study aims to evaluate the diagnostic performance of DNA methylation biomarkers in detecting urothelial carcinoma in patients with hematuria. By collecting preoperative urine samples from a small cohort of hematuria patients and performing DNA methylation testing, we aim to explore the feasibility and advantages of this method in clinical applications.
3. Methods

   Study Design:

   This is a prospective pilot study aimed at evaluating the effectiveness of DNA methylation biomarkers in detecting urothelial carcinoma in patients with hematuria.

   Sample Size Calculation:

   Based on our previous observations, the incidence of urothelial carcinoma in patients with hematuria is 20%-30%, slightly higher than reported in other literature. Therefore, we hypothesize that 25% of the patients in the hematuria cohort have UC. The group allocation ratio (R): N-/N+ = 75%/25% = 3.

   Assumptions:

   Area under the curve (AUC) under H0: 0.5 AUC under H1: 0.8 Power: 0.95 Significance level (Alpha): 0.05 Type of data: Continuous FPR range: 0.00 to 1.00

   Results: Using PASS 15.0 software for sample size calculation to ensure sufficient statistical power. The calculated sample size is:

   N+ (number of patients with UC): 14 N- (number of patients without UC): 42 Total sample size (N): 56

   Considering a 20% dropout rate, the adjusted sample size is:

   N+': 18 N-': 53 Total sample size (N'): 71

   Inclusion and Exclusion Criteria:

   Inclusion Criteria:

   Aged between 18 and 99 years, with gross or microscopic hematuria (>3/HP). Able to provide 50ml urine for testing before surgery. Consent to participate in the study and sign the informed consent form.

   Exclusion Criteria:

   With history of malignancy or concomitant malignancies other than UC. Severe urinary tract infection leading to sepsis. Patients with indwelling catheters, nephrostomy, or cystostomy. Severe liver or kidney failure or other conditions deemed unsuitable for the study.

   Patients who did not undergo surgical treatment for various reasons. Samples with insufficient DNA content or other quality control failures.

   Sample Collection:

   Clinicians will collect fresh urine samples from enrolled hematuria patients and record their basic information, clinical information, and medical history.

   Samples will be randomly numbered and provided to DNA methylation testing personnel to ensure blinding.

   Testing Method:

   Urine samples were collected in EP Genomic DNA Kit with an automated nucleic acid extraction instrument. Subsequently, 100 ng of genomic DNA was used for methylation-sensitive restriction enzyme qPCR (MSRE-qPCR) detection as described previously. Different from bisulfite PCR relying on bisulfite conversion, MSRE-qPCR is based on the selective digestion of DNA by methylation-sensitive enzyme followed by qPCR with primers that surround the cutting site.

   Unblinding and Data Organization:

   After the last sample is successfully enrolled and tested, non-recruiting personnel and testing personnel will unblind the samples and organize clinical and pathological information.

   Data Analysis:

   Using pathological results as the gold standard. Calculate the sensitivity, specificity, positive predictive value, and negative predictive value of DNA methylation biomarkers.

   Use statistical methods (such as ROC curves) to evaluate the diagnostic performance of DNA methylation biomarkers and calculate the AUROC.

   Ethics and Informed Consent:

   This study has been approved by the hospital's ethics committee, and all participants must sign an informed consent form.
4. Conclusion This study aims to validate the effectiveness of urine DNA methylation testing in detecting urothelial carcinoma in patients with hematuria and provide evidence for its clinical application. The results of this preliminary study will offer essential data support and design optimization suggestions for future larger-scale studies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 99 years, with gross or microscopic hematuria (>3/HP).
2. Able to provide 50ml urine for testing before surgery.
3. Consent to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. With history of malignancy or concomitant malignancies other than UC.
2. Severe urinary tract infection leading to sepsis.
3. Patients with indwelling catheters, nephrostomy, or cystostomy. 4 Severe liver or kidney failure or other conditions deemed unsuitable for the study.

5. Patients who did not undergo surgical treatment for various reasons. 6. Samples with insufficient DNA content or other quality control failures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective pilot study aimed at evaluating the effectiveness of DNA methylation biomarkers in detecting urothelial carcinoma in patients with hematuria.
Sampling Method: Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of DNA methylation test | 1 year
  Evaluate the diagnostic performance of DNA methylation biomarkers by calculating the AUROC value.

SECONDARY OUTCOMES:
Sensitivity, specificity, positive predictive value, and negative predictive value of DNA methylation biomarkers | 1 year
  Calculate the sensitivity, specificity, positive predictive value, and negative predictive value of DNA methylation biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China